CLINICAL TRIAL: NCT00800644
Title: Evaluation of Bone Density and Pelvic Fractures in Women Undergoing Definitive Pelvic Radiation Therapy for Cervical, Endometrial or Vaginal Cancer
Brief Title: Pelvic Fractures and Radiation Therapy for Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0023
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Cervical Cancer; Endometrial Cancer; Vaginal Cancer
Keywords: Cervical Cancer; Endometrial Cancer; Vaginal Cancer; Cervix; Endometrial; X-ray; Computed tomography; Magnetic resonance imaging; Vagina; Pelvic radiation therapy; Bone density; Bone mineral density test; Pelvic fractures; Gynecologic Oncology; Bone turnover
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Vaginal Neoplasms; Hip Fractures | interventions — Magnetic Resonance Spectroscopy; Hematologic Tests; X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Evaluation Group: Bone Mineral Density Test + MRI or CT + Blood Test
  Interventions: Procedure: CT or MRI + Blood Test

INTERVENTIONS:
Procedure: CT or MRI + Blood Test — During routine visits, a magnetic resonance imaging (MRI) scan or a computed tomography (CT) scan.
  Blood (about 1 tablespoon) will be drawn to test for bone turnover.
  Other Names: x-ray; computed tomography; magnetic resonance imaging

SUMMARY:
The goal of this study is to estimate how often pelvic fractures occur in women treated with radiation therapy for either newly diagnosed or recurrent cervical, endometrial, or vaginal cancer. The study will also estimate the changes in bone mineral density and the changes in the blood that relate to "bone turnover". High bone turnover can weaken bones and make you more likely to break a bone.

DETAILED DESCRIPTION:
If you agree to take part in this study, the following tests and procedures will be performed before radiation therapy:

* You will have a bone mineral density test. A bone mineral density test measures bone loss over time, identifies osteoporosis (a disease of the bones that causes them to be weak and easily breakable) or the risk for developing osteoporosis, and checks your risk for fractures. During the test, you will lie on a cushioned table while a mechanical arm-like device will pass over your body. This device will not touch you.
* During your routine visits, you may have either a magnetic resonance imaging (MRI) scan or a computed tomography (CT) scan of the pelvis as part of your standard of care. A PET scan may be done if your doctor thinks it is necessary. These scans will be reviewed by the research staff of this study to determine your response to therapy, determine if your cancer has returned, and to look for broken bones.
* Blood (about 1 tablespoon) will be drawn to test for bone turnover.
* Blood (about 2 to 3 teaspoons) will be drawn for tests to measure the level of vitamin D, calcium, phosphorus, and parathyroid hormone (PTH).
* Researchers will collect information from your medical record. This information will include your medical history, your ethnicity, if you have had any bone fractures, if you have a history of bone fractures in your family, and your use of tobacco and/or alcohol.

At 4 weeks after start of radiation therapy, blood (about 2 to 3 teaspoons) will be drawn to test for bone turnover.

At 3 months, 1 year, and 2 years after you complete radiation:

* You will have a bone mineral density test.
* You may have either an MRI or CT scan of the pelvis as part of your standard of care. A PET scan may be done if your doctor thinks it is necessary. These scans will be reviewed by the research staff of this study to determine your response to therapy, determine if your cancer has returned, and to look for broken bones.
* Blood (about 2 tablespoons) will be drawn for tests to measure the level of vitamin D and to test for bone turnover.

Length of Study:

You will be off study 2 years after you complete radiation.

After 2 years and for up to 5 years, results of bone density tests or scans of the pelvis that you have outside of this study will be collected.

This is an investigational study.

Up to 300 women will take part in the study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed primary or recurrent cervical , endometrial or vaginal cancer. All stages, grades and histologic subtypes will be eligible except neuroendocrine.
2. Patients treated with definitive radiation therapy. Patients receiving extended field radiation or brachytherapy in addition to pelvic radiation are eligible. Patients treated with surgery, chemotherapy and/or hormonal therapy in addition to radiation therapy are also eligible.
3. Patients must sign an approved informed consent document.

Exclusion Criteria:

1. Patients undergoing palliative intent radiation therapy for advanced disease.
2. Patients who received prior radiation to the pelvis.
3. Patients with an existing pelvic fracture within the proposed radiation field.
4. Patients unwilling or unable to provide informed consent for the study.
5. Patients with bone metastases.
6. Neuroendocrine features present.
7. Patients weighing more than 300 lbs are excluded as they cannot be adequately studied in axial skeleton with current bone mineral density software.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cervical, endometrial, or vaginal cancer patients who will receive extended field radiation, brachytherapy, or pelvic radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2008-11-05 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Bone Mineral Density (BMD) | 2 years

SECONDARY OUTCOMES:
Incidence of pelvic fractures incidence in women treated with definitive pelvic radiation therapy for cervical, endometrial or vaginal cancer | Within 2 years of treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Schmeler, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Salcedo MP, Sood AK, Jhingran A, Eifel PJ, Klopp AH, Iyer RB, Fellman BM, Jimenez C, Schmeler KM. Pelvic fractures and changes in bone mineral density after radiotherapy for cervical, endometrial, and vaginal cancer: A prospective study of 239 women. Cancer. 2020 Jun 1;126(11):2607-2613. doi: 10.1002/cncr.32807. Epub 2020 Mar 3. PMID 32125711
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org